CLINICAL TRIAL: NCT06643845
Title: Is Non Surgical CaRE Using Treat to Target Multimodal meDIcal Strategies aBLE to Delay or Avoid Total Knee Replacement? (INCREDIBLE)
Brief Title: Can Multimodal Medical Strategies Can Delay Total Knee Replacement?
Acronym: INCREDIBLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29BRC23.0002
Record Dates: First submitted 2024-08-19; First posted 2024-10-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Surgery; Arthroplasty; Total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal medical care arm (Experimental): In the medical care arm, rheumatologists will list previous treatment, ongoing treatment and then order validated treatment (corticosteroid or hyaluronic acid joint injection if necessary, physical activity and weight loss in the event of obesity, other non-drug treatments (insole, orthosis) as well as other drug treatments (pain killers or non steroidal anti-inflammatory drugs) including validated tools (personalized program, filmed sessions and digital exercise media for regular practice at home, motivational e-mails). At least one modification will be discussed in each domain (physical activity, weight loss, insole, orthosis, assistive device when walking, joint injection, pills -pain killer acetaminophen and opioids- nonsteroidal anti inflammatory drugs -with classical rules - and others)
  Interventions: Other: Medical and non-medical treatments
- Surgery arm (Active Comparator): In the surgery arm, patients will have to plan, as initially suggested, their surgery (total knee arthroplasty)
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthroplasty — In the surgery arm, patients will have their surgery (arthroplasty), as originally planned.
  Arms: Surgery arm
Other: Medical and non-medical treatments — In the medical care arm, patients will follow multimodal medical strategies to prevent surgery in a population of patients with knee osteoarthritis having a first indication of knee prosthesis
  Arms: Multimodal medical care arm

SUMMARY:
Knee is the most common site of osteoarthritis. Treatment of knee osteoarthritis starts with a full course of medical therapy, followed by surgery to replace the knee with a prosthesis if this strategy fails, or in advanced cases. However, the new recommendations of the French rheumatology society, which evaluate the various treatments and position them in the treatment plan, are not well known, and the definition of a complete treatment remains unclear. The vast majority of patients are therefore referred to a surgeon after having tried a small part of the therapeutic arsenal (generally analgesics and corticosteroid or hyaluronic acid infiltrations). The goal of this study is to to select patients most likely to gain from surgery and to develop strategies that avoid the need for major surgery.

DETAILED DESCRIPTION:
Knee is the most common site of osteoarthritis. Treatment of knee osteoarthritis starts with a full course of medical therapy, followed by surgery to replace the knee with a prosthesis if this strategy fails, or in advanced cases.

However, the new recommendations of the French rheumatology society, which evaluate the various treatments and position them in the treatment plan, are not well known, and the definition of a complete treatment remains unclear. The vast majority of patients are therefore referred to a surgeon after having tried a small part of the therapeutic arsenal (generally analgesics and corticosteroid or hyaluronic acid infiltrations).

Yet medical treatment has proved effective, suggesting that it could prevent a significant number of total knee arthroplasties. In addition, osteoarthritis of the knee is associated with various co-morbidities (diabetes, cardiovascular) that medical treatment can minimize (diet, physical activity).

The effectiveness of knee prostheses has been demonstrated, but up to 20% of patients continue to experience pain, and surgical procedures induce rare but serious events. Prostheses can also be revised, and are expensive.

This research is designed for patients suffering from femoro-tibial osteoarthritis who have been proposed total knee replacement by a surgeon, and aims to develop strategies to avoid the need for major surgery until the medical treatment arsenal adapted to the patient's situation has been tried.

In the treatment of osteoarthritis, the impact of shared decision-making between rheumatologists, orthopaedic surgeons and the patient in the event of incomplete medical treatment has been shown to be important, as the decision is often modified after discussion.

The main objective of this prospective, randomized, pragmatic, non-blinded, multicenter study is to investigate whether shared decision-making coupled with multimodal medical strategies delays surgery by at least 2 years in most patients, with non-inferiority on pain and function, lower cost and fewer serious adverse events compared with total knee arthroplasty from the outset.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years old
* Femoro-tibial osteoarthritis Kellgren stage stage≥ 2 without laxity in extension;
* A proposal of total knee replacement by a surgeon;
* No corticosteroid joint injection within 3 months;
* Visual analogic score pain (VAS) >40/100 but <90/100 or Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index function sub scale >40/100 at inclusion;
* Wish to discuss medical care;
* Able to consent and having signed a consent form.

Exclusion Criteria:

* Contraindication or no indication to surgery or medical care (severe infection for example)
* Inflammatory arthritis
* Lack of social insurance
* Symptomatic (VAS pain >40) contralateral knee or hip osteoarthritis (with or without replacement)
* Pregnant or breastfeeding woman
* Patient under court protection, guardianship, curatorship
* Patient deprived of liberty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Multimodal medical care osteoarthritis is non inferior (with a threshold of 15% for pain and function) to total knee arthroplasty in symptomatic radiographic knee osteoarthritis. | 2 years
  The outcome relates to two scales which constitute the composite principal endpoint;
  * Visual Analogic Score pain, VAS (scale 0-100)
  * Western Ontario and McMaster Universities function, WOMAC (scale 0-100) Success is defined by a VAS AND WOMAC scale ≤40/100 at 2 years Failure is defined by a VAS pain OR WOMAC scale > 40/100 at 2 years.

SECONDARY OUTCOMES:
Study the proportion of delayed surgery in the medical group | 2 years
  Number of cumulated surgery (yes/no) by month in the medical group
Study the proportion of patients with severe events induced by surgery | 2 years
  Number of severe events (Who classification) in the surgical group.
Analyze the impact of physical activity on change of body mass by arm in the randomized population. | 2 years
  Perform analyses of body mass on whole body densitometry
To compare analgesic use by arm. | 2 years
  Analgesic use by class in milligram.
To compare the 0-2 years cost using the National Health Data System between the 2 groups. | 0-2 years
  Cost in euro between 0-2
To compare the 2-5 cost using the National Health Data System between the 2 groups. | 2-5 years
  Cost in euro between 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alain Saraux, Pr, Principal Investigator — CHU Brest
Locations (21):
- France (21):
  - CHU Amiens, Amiens
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHD Vendée, La Roche-sur-Yon
  - CHU Le Mans, Le Mans
  - CHU Limoges, Limoges
  - GHICL- Hôpital Saint Philibert, Lomme
  - HCL, Lyon
  - CHU Montpellier, Montpellier
  - CH Morlaix, Morlaix
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - AP-HP Cochin, Paris
  - AP-HP La pitié, Paris
  - AP-HP Lariboisière, Paris
  - AP-HP Saint-Antoine, Paris
  - CHIC Quimper, Quimper
  - CHU Reims, Reims
  - CHU Saint Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access request will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.